CLINICAL TRIAL: NCT01228981
Title: Observational Study to Assess Genotypes/Phenotypes Correlations in Type-2 Diabetic Retinopathy
Acronym: CEC120
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Collaborators: University of Coimbra (Other)
Responsible Party: Sponsor
Other Study IDs: PTDC/SAU-OSM/103226/2008
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Type-2 Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type-2 Diabetic Retinopathy

SUMMARY:
The purpose of this study is to characterize type 2 diabetic patients with initial alterations of diabetic retinopathy (DR) based on 3 different phenotypes previously identified and different patterns of progression in order to correlate this data with genetic information.

DETAILED DESCRIPTION:
This study aims to to characterize type 2 diabetic patients with initial alterations of diabetic retinopathy (DR) based on three different phenotypes previously identified and different patterns of progression [Lobo, 2004] in order to correlate this data with genetic information (based on a list of candidate genes previously identified as being involved in DR).

The results of this study will be used exclusively for scientific purposes.

ELIGIBILITY:
Inclusion Criteria:

* Type-2 diabetic subjects form the PTDC/SAU-OSM/72635/2006 clinical trial (early stages of non-proliferative retinopathy - level 30 to 35 ETDRS;. females or males; age over 18 years) with a signed Informed Consent for this study.

Exclusion Criteria:

* Cataract or other eye disease that may interfere with fundus examinations; Vitreous syneresis or posterior vitreous detachment; and Dilatation of the pupil < 5 mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type-2 diabetic subjects in the early stages of non-proliferative retinopathy (level 30 to 35 ETDRS) included in the clinical trial "Validation of a predictive model to estimate the risk of conversion to clinically significant macular edema and/or vision loss in mild nonproliferative diabetic retinopathy in diabetes type 2" (Protocol number: PTDC/SAU-OSM/72635/2006; ongoing at AIBILI Clinical Trial Center).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Phenotypes of Diabetic Retinopathy progression. | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Lobo, MD PhD, Principal Investigator — Association for Innovation and Biomedical Research on Light and Image
Locations (1):
- AIBILI - Clinical Trials Center, Coimbra, Coimbra District, Portugal

REFERENCES:
- [Derived] Cunha-Vaz J, Ribeiro L, Lobo C. Phenotypes and biomarkers of diabetic retinopathy. Prog Retin Eye Res. 2014 Jul;41:90-111. doi: 10.1016/j.preteyeres.2014.03.003. Epub 2014 Mar 26. PMID 24680929
- See also: Related Info — http://www.aibili.pt